CLINICAL TRIAL: NCT02548104
Title: Randomized, Double-Blinded Study to Evaluate the Analgesic Efficacy of Anterior Femoral Cutaneous Nerve Block and/or Genicular Nerve Block When Combined With Adductor Canal (Saphenous) Nerve Block After Total Knee Arthroplasty
Brief Title: Analgesic Efficacy of Anterior Femoral, Genicular and Adductor Canal Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Jun Tang, MD, Department of anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSMCPro00034213; NCT02167282 (obsolete NCT alias)
Record Dates: First submitted 2015-09-08; First posted 2015-09-14 (Estimated); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor canal block (ACB) (Active Comparator): Group I Adductor canal block (ACB): 0.25% bupivacaine with 1:200,000 epinephrine 30 ml and ultrasound-guided genicular (IPACK) with normal saline 15 ml
  Interventions: Other: ACB
- Adductor canal ACB + genicular (IPACK) (Experimental): Group II Adductor canal block (ACB): 0.25% bupivacaine with 1:200,000 epinephrine 30 ml and ultrasound-guided genicular (IPACK) with 0.25% Bupivicaine with 1:200,000 epinephrine 15 ml
  Interventions: Other: ACB + iPACK

INTERVENTIONS:
Other: ACB — ultrasound-guided ACB with 0.25% Bupivicaine with 1:200,000 epinephrine 30 ml and ultrasound-guided genicular (IPACK) with normal saline 15 ml
  Arms: Adductor canal block (ACB)
Other: ACB + iPACK — ultrasound-guided ACB with 0.25% Bupivicaine with 1:200,000 epinephrine 30 ml and ultrasound-guided genicular (IPACK) with 0.25% Bupivicaine with 1:200,000 epinephrine 15 ml
  Arms: Adductor canal ACB + genicular (IPACK)

SUMMARY:
Recently, more distal approach to femoral nerve branches (saphenous) in the adductor canal in the medial compartment of the thigh have shown to provide comparable anesthesia and analgesia without quadriceps muscle weakness than traditional femoral nerve blocks (FNB) after total knee arthroplasty (TKA). Adductor canal block (ACB) has the unique advantage of providing localized analgesia to the peripatellar and intra-articular aspects of the knee joint without reducing the patient's ability to perform a straight leg raise. However, it does not adequately address the incisional pain component on the anterior surface of the knee innervated by anterior femoral cutaneous nerve. This pain may be improved by addition of the anterior femoral block (AFB). Additionally, the ACB does not provide analgesia to the posterior aspect of the knee, which is commonly moderate to severe after surgery. This pain may be decreased by addition of the genicular block, also known as the iPACK block (interspace between the popliteal artery and the capsule of the knee). There is no study that has evaluated the potentially analgesic benefits of the AFB or the iPACK block combined with ACB after TKA. Therefore, the investigators designed this randomized, prospective, and double-blinded study to assess our hypothesis that the addition of the AFB and/or iPACK block to the ACB will improve analgesic effects, decrease pain scores, deceased opioid requirement, and as well as facilitate early recovery and improve patient satisfaction with pain management in patient after TKA.

DETAILED DESCRIPTION:
Postoperative pain associated with total knee arthroplasty (TKA) can pose significant challenges in the recovery process of the patients undergoing this procedure. Traditionally, opioids have played a significant role in treating postoperative pain. It is well established that opioids are highly effective in relieving pain at rest, but are less effective in relieving pain associated with motion (e.g. ambulation, passive motion, and physical rehabilitation). Furthermore, the use of opioids for analgesia is associated with well-known side effects (such as: nausea, vomiting, constipation, ileus, bladder dysfunction, respiratory depression, pruritus, drowsiness, sedation, and allergic reaction). These opioid side effects, which range in severity, can significantly interfere with the rehabilitation process and contribute to a delay in hospital discharge.

Significant interest exists in the application of regional anesthetic techniques as an adjuvant to traditional opioid analgesics for pain control in patients after TKA. Specifically, the incorporation of femoral nerve blocks (FNB) as an adjunct in postoperative pain control has been widely reported in the anesthesia literature. While it has shown to be effective in post-operative pain control, it has introduced additional challenges for physical therapy and raised new concerns regarding the associated quadriceps muscle weakness. Until adequate quadriceps function returns, the need for knee immobilization devices to protect patients with traditional FNB from falls interferes with the early recovery process and the achievement of physical therapy milestones.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-90 yrs
2. The American Society of Anesthesiologists (ASA) Physical Status 1-3
3. Either gender

Exclusion Criteria:

1. Refusal to participate in the study
2. Age< 18 yrs, or> 90 yrs
3. General anesthesia
4. Bilateral TKA, or revision of TKA
5. Contraindications to regional blockage including but not limited to:

   * Patient refusal to regional blockade
   * Infection at the site of needle insertion
   * Systemic infection
   * Bleeding diathesis or coagulopathy (as diagnosed by history or laboratory evaluation)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Changes of pain scores (VRS) at rest | Post-op day 1,2,3
  Verbal rating scale (VRS) scores: 0 = none to 10 = intolerable pain.
Changes of pain scores (VRS) at motion activity | Post-op day 1,2,3
  Verbal rating scale (VRS) scores: 0 = none to 10 = intolerable pain.

SECONDARY OUTCOMES:
Patient satisfaction score | Post-op day 1
  (0-very dissatisfied to 10 very satisfied)
Patient satisfaction score | Post-op day 2
  (0-very dissatisfied to 10 very satisfied)
Patient satisfaction score | Post-op day 3
  (0-very dissatisfied to 10 very satisfied)
Gait distance | Post-op day 1
  (feet)
Gait distance | Post-op day 2
  (feet)
Gait distance | Post-op day 3
  (feet)

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, M.D.,PhD., Principal Investigator — Department of Anesthesiology
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States